CLINICAL TRIAL: NCT04849650
Title: An Open Label Study of the Pharmacokinetics of Intravenous and Oral Amisulpride in Adults With Severe Renal Impairment and Healthy Control Subjects
Brief Title: PK Study of IV and Oral Amisulpride in Subjects With Severe Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acacia Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DP10026
Record Dates: First submitted 2021-04-14; First posted 2021-04-19 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Renal Disease, End Stage
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Amisulpride

STUDY DESIGN:
Intervention Model Description: One group of subjects with renal impairment will receive 10mg IV Amisulpride followed 24 hours later by a 10mg oral dose.
  One group of matched healthy subjects will receive 10mg IV Amisulpride followed 24 hours later by a 10mg oral dose.
Masking Description: All parties will have knowledge of the interventions assigned to each subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Renal Impairment Subjects (Experimental): 10mg dose of IV Amisulpride, followed 24 hours by a 10mg oral dose of Amisulpride
  Interventions: Drug: Amisulpride IV; Drug: Amisulpride Oral Tablet
- Healthy Subjects (Experimental): 10mg dose of IV Amisulpride, followed 24 hours by a 10mg oral dose of Amisulpride
  Interventions: Drug: Amisulpride IV; Drug: Amisulpride Oral Tablet

INTERVENTIONS:
Drug: Amisulpride IV — A single 10mg IV dose of Amisulpride given over 1 minute
Drug: Amisulpride Oral Tablet — A single 10mg dose given as an oral tablet

SUMMARY:
The aim of the study is to understand how Amisulpride is taken up and distributed around the body and how quickly it is eliminated, when given by mouth and into a vein in adults with severe kidney disease. In addition it is important to understand how well tolerated Amisulpride is in this patient population. Healthy adults will be studied to provide a comparison.

DETAILED DESCRIPTION:
This will be an open-label, non-randomised, pharmacokinetic study in

* 6 adult subjects with severe renal impairment and end-stage renal disease (i.e., eGFR < 30 mL/min/1.73 m2) without dialysis.
* 6 matched healthy subjects (control group).

Each subject will be given a single dose of 10 mg IV Amisulpride, followed by a single dose of 10 mg oral Amisulpride given 24 hours later.

Subjects will be admitted to the clinic on Day -1. Dosing will start the following day (Day 1). Serial blood samples will be taken during Days 1-3 to assess the pharmacokinetics of Amisulpride. Subjects will remain in clinic over the duration of the study and will be discharged when the final blood sample is drawn on Day 3.

The tolerability /safety of Amisulpride will be assessed by clinical chemistry and haematology assessments, vital signs, electrocardiograms (ECG), physical examination and adverse event reporting.

ELIGIBILITY:
Inclusion Criteria: Healthy Subjects

1. Age 18 to 75 years of age at time of signing ICF.
2. Body mass index (BMI) between 18 and 38 kg/m2.
3. Must be willing and able to communicate and participate in the whole study.
4. Must provide written informed consent.
5. Must agree to use an adequate method of contraception
6. Healthy as defined by:

   * The absence of clinically significant illness and surgery within 4 weeks prior to dosing. Subjects vomiting within 24 hours pre-dose will be carefully evaluated for upcoming illness/disease. Inclusion pre-dosing is at the discretion of the Principal Investigator;
   * The absence of clinically significant history of neurological, endocrine, cardiovascular, pulmonary, hematological, immunologic, psychiatric, gastrointestinal, renal, hepatic (including cholecystectomy), and metabolic disease;
   * The absence of clinically significant history of lactic acidosis and severe hepatomegaly with steatosis;
   * The absence of history of suicidal tendency, disposition to seizures, state of confusion, or clinically relevant psychiatric diseases.
7. Normal renal function, i.e., eGFR or creatinine clearance ≥ 90 mL/min/1.73 m2 as calculated using the MDRD4 or Cockcroft-Gault equation; at the Principal Investigator's discretion, 24 hour creatinine clearance may be conducted to determine renal function.
8. Matched to subjects with severe renal impairment for gender, age (± 10 years), and BMI (± 15%) to the extent possible.

Inclusion Criteria: Renal Impaired Subjects

1. Age 18 to 75 years of age at time of signing ICF.
2. Body mass index (BMI) between 18 and 38 kg/m2.
3. Must be willing and able to communicate and participate in the whole study.
4. Must provide written informed consent.
5. Must agree to use an adequate method of contraception
6. A diagnosis of renal impairment that has been stable, without significant change in overall disease status in the 3 months prior to screening as determined by the Principal Investigator, with no requirement for dialysis, and an eGFR at screening < 30 mL/min/1.73 m2 calculated using the MDRD4 equation.

Exclusion Criteria: Healthy Subjects

1. Subjects who have received any IMP in a clinical research study within the 30 days prior to IMP administration on this study.
2. Subjects who are study site, CRO or sponsor employees, or immediate family members of a study site, CRO or sponsor employee.
3. Subjects who have previously been enrolled in this study.
4. Women who are pregnant or breastfeeding.
5. Subjects who have received amisulpride for any indication within the 30 days prior to dosing.
6. Allergy to amisulpride or any of the excipients of amisulpride.
7. History of any drug or alcohol abuse in the 2 years prior to screening.
8. Regular alcohol consumption >21 units per week in the 6 months prior to screening.
9. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening.
10. History of epilepsy in the 5years prior toscreening.
11. History of clinically significant syncope.
12. Family history of sudden death.
13. Family history of premature cardiovascular death.
14. Clinically significant history or family history of congenital long QT syndrome (e.g.

    Romano-Ward syndrome, Jervell and Lange-Nielson syndrome) or Brugada's syndrome.
15. History of clinically significant arrhythmias or ischaemic heart disease (especially ventricular arrhythmias, atrial fibrillation (AF), recent conversion from AF or coronary spasm).
16. Conditions predisposing the volunteer to electrolyte imbalances (e.g. altered nutritional states, chronic vomiting, anorexia nervosa, bulimia nervosa).
17. Clinically significant abnormal biochemistry,haematology or urinalysis at screening as judged by the investigator
18. Positive drugs of abuse test result
19. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results at screening.
20. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening or menses) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the dosing.
21. Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than 2,000 mg per day acetaminophen) or herbal remedies in the 14 days before IMP administration
22. Administration of a biological product in the context of a clinical research study within 90 days prior to dosing, or concomitant participation in an investigational study involving no drug or device administration.
23. Failure to satisfy the investigator of fitness to participate for any other reason.

Exclusion Criteria: Renal Impaired Subjects

1. Subjects who have received any IMP in a clinical research study within the 30 days prior to IMP administration on this study.
2. Subjects who are study site, CRO or sponsor employees, or immediate family members of a study site, CRO or sponsor employee.
3. Subjects who have previously been enrolled in this study.
4. Women who are pregnant or breastfeeding.
5. Subjects who have received amisulpride for any indication within the 30 days prior to dosing.
6. Allergy to amisulpride or any of the excipients of amisulpride.
7. History of any drug or alcohol abuse in the 2 years prior to screening.
8. Regular alcohol consumption >21 units per week in the 6 months prior to screening.
9. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening.
10. History of epilepsy in the 5years prior to screening.
11. History of clinically significant syncope.
12. Family history of sudden death.
13. Family history of premature cardiovascular death.
14. Clinically significant history or family history of congenital long QT syndrome (e.g.

    Romano-Ward syndrome, Jervell and Lange-Nielson syndrome) or Brugada's syndrome.
15. History of clinically significant arrhythmias or unstable ischaemic heart disease (especially ventricular arrhythmias, atrial fibrillation (AF), recent conversion from AF or coronary spasm).
16. Positive drugs of abuse test result, unless caused by a documented prescription drug.
17. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results at screening.
18. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening or menses) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the dosing.
19. Administration of a biological product in the context of a clinical research study within 90 days prior to dosing, or concomitant participation in an investigational study involving no drug or device administration.
20. Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
PK: Amisulpride plasma exposure (AUC) after a single IV dose | 24 hours
  Amisulpride plasma exposure after a single IV dose measured as the area under the concentration-time curve (AUC) between study drug administration and the time at which the following-day oral dose of Amisulpride is given

SECONDARY OUTCOMES:
PK: Amisulpride plasma exposure (AUC) after a single oral dose | 24 hours
  Amisulpride plasma exposure after a single oral dose measured as the area under the concentration-time curve (AUC) from study drug administration extrapolated to infinity
PK: Cmax | 24 hours
  Peak plasma concentration (Cmax), for both a single IV and single oral dose.
PK: Tmax | 24 hours
  Time at which peak plasma concentration achieved (Tmax) for both a single IV and single oral dose.
PK: T1/2 | 24 hours
  Half-life (T1⁄2) of both a single IV and single oral dose.
PK: Clearance | 24 hours
  Clearance of both a single IV and single oral dose.
PK: Vd | 24 hours
  Volume of distribution (Vd) of both a single IV and single oral dose.
Safety: AE | From first study drug administration until discharge (4 days)
  Frequency and severity of treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Fox, MD, Study Director — Chief Medical Officer
Locations (1):
- Panax Clinical Research, Miami Lakes, Florida, United States

IPD SHARING:
Plan to Share IPD: No